CLINICAL TRIAL: NCT06644352
Title: A Prospective, Randomized, Controlled, Multicenter Study Comparing the Right Versus Left Thoracic Surgical Approaches for Locally Advanced Siewert II Gastroesophageal Junction Adenocarcinoma After Neoadjuvant Chemotherapy
Brief Title: Right Versus Left Thoracic Surgical Approaches for Siewert II Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YLI
Record Dates: First submitted 2024-07-12; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Siewert Type II Adenocarcinoma of Esophagogastric Junction
Keywords: GastroEsophageal Cancer; Surgical Incision; Left thoracic incision; Right thoracic incision; Neoadjuvant chemotherapy
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right thoracic approach (Experimental): Neoadjuvant therapy+surgery+adjuvant therapy. Neoadjuvant therapy: chemotherapy with 2-4 cycles； Surgery: dissociate the stomach and operate the gastroesophagostomy and lower mediastinal lymphadenectomy by the right thoracic approach (right thoracic incision); Adjuvant therapy: perioperative chemotherapy with total 8 cycles (including neoadjuvant chemotherapy).
  Interventions: Procedure: different thoracic surgical approaches
- Left thoracic approach (Active Comparator): Neoadjuvant therapy+surgery+adjuvant therapy. Neoadjuvant therapy: chemotherapy with 2-4 cycles； Surgery: dissociate the stomach and operate the gastroesophagostomy and lower mediastinal lymphadenectomy by the left thoracic approach (including right thoracic and abdominal incision); Adjuvant therapy: perioperative chemotherapy with total 8 cycles (including neoadjuvant chemotherapy).
  Interventions: Procedure: different thoracic surgical approaches

INTERVENTIONS:
Procedure: different thoracic surgical approaches — Right Versus Left Thoracic Surgical Approaches

SUMMARY:
To explore the 5-year overall survival (OS) of right versus left thoracic surgical approaches for patients with locally advanced Siewert II gastroesophageal junction adenocarcinoma treated by neoadjuvant chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed gastroesophageal adenocarcinoma;
2. R0 resectable Siewert Ⅱ, cT2-3N0-3M0 (AJCC V8 TNM classification);
3. Have a performance status of 0 or 1 on the ECOG Performance Scale;
4. Age 18-80 years old, both men and women;
5. Estimated survival ≥6 months;
6. Be willing and able to provide written informed consent/assent for the trial;
7. Demonstrate adequate organ function ;
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 7 days before enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;
9. Have not received systemic or local treatment for esophageal cancer in the past.

Exclusion Criteria:

1. Have a history of other malignant tumors in the past or at the same time;
2. Previous upper abdominal surgery (excluding cholecystectomy);
3. Bleeding, perforation and obstruction requiring emergency surgical treatment;
4. Severe heart, lung, liver and kidney dysfunction, which the researcher thinks is not suitable for operation;
5. Hydrothorax and ascites with clinical symptoms need therapeutic puncture or drainage;
6. Participate in other clinical studies or less than 1 month from the end of the previous clinical study;
7. Have a history of psychoactive drug abuse, alcoholism or drug abuse;
8. Be unable or do not agree to bear the inspection and treatment expenses at their own expense;
9. The researcher thinks that it should be excluded from this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
OS rate | 5 years
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
DFS rate | 3 years
  DFS is defined as the time from randomization to the first documented disease progression of local recurrence or distant metastasis or death due to any cause.
pCR rate | 1 month after resection
  PCR is defined as pT0N0M0
MPR rate | 1 month after resection
  MPR is defined as viable tumor comprised ≤ 10% of resected tumor specimens.
Operative Complications | perioperative period
  Operative Complications

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China